CLINICAL TRIAL: NCT03239665
Title: Randomized Trial of Peer-to-Peer Versus Pharmacist Education to Improve Older Adults' Vaccination Knowledge Through the Senior Center Model of Care
Brief Title: Vaccination Education Through Pharmacists and Senior Centers (VEPSC)
Acronym: VEPSC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Thomas Jefferson University (Other)
Responsible Party: Principal Investigator, Laura T. Pizzi, PharmD, MPH, Professor and Director, Center for Health Outcomes, Policy, & Economics, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro20170000208
Record Dates: First submitted 2017-07-20; First posted 2017-08-04 (Actual); Results first posted 2020-07-01 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Infectious Disease; Pneumonia, Bacterial; Influenza; Zoster; Herpes
Keywords: Vaccine; Educational intervention; Senior Center Model of Care; Older adults
MeSH Terms: conditions — Communicable Diseases; Pneumonia, Bacterial; Influenza, Human; Chickenpox

STUDY DESIGN:
Intervention Model Description: The design is a randomized trial with randomization to PHARM or PEER performed at the program date level.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pharmacist-led Intervention (PHARM) (Active Comparator): In the PHARM intervention group, participants will be given a 60-minute formal presentation on vaccine-preventable diseases to address knowledge and beliefs related to zoster, pneumonia, and influenza and to address barriers to receiving vaccination. In several studies, it has been demonstrated that those who believe it is wise to receive vaccinations and those that have discussed vaccination with their healthcare provider are more likely to receive a vaccine.
  Interventions: Behavioral: Pharmacist-led Intervention (PHARM)
- Peer-led Intervention (PEER) (Experimental): A pharmacist will train the peer educators about vaccine-preventable diseases over the course of two didactic sessions. Following this training, a third session will be held to train the peer educators on the script that they will deliver to participants. The script will include the key learning points to be taught by the peer educators to participants about vaccine preventable diseases and vaccination. The script will also include role-play exercises. In the role-play exercises, 3 vaccination-related scenarios (one for each disease- zoster, pneumonia, and influenza) will be delivered to illustrate situations participants might encounter when interacting with healthcare providers or friends/family.
  Interventions: Behavioral: Peer-led Intervention (PEER)

INTERVENTIONS:
Behavioral: Pharmacist-led Intervention (PHARM) — 60 minute didactic lecture about vaccinations.
  Arms: Pharmacist-led Intervention (PHARM)
Behavioral: Peer-led Intervention (PEER) — 60 minute peer led small group intervention including skits and other educational material
  Arms: Peer-led Intervention (PEER)

SUMMARY:
The study consists of two arms (PHARM and PEER) designed to educate participants about three vaccine-preventable diseases (zoster, pneumonia, and influenza) and vaccination. PHARM will consist of a 60-minute presentation about the three vaccine-preventable diseases and their vaccinations delivered by a pharmacist, featuring a didactic lecture and discussion supplemented by video clips of community members discussing their experiences around vaccination, as well as physicians underscoring the importance of vaccination. PEER will consist of a 60-minute small-group session led by a peer educator which includes scripted roleplaying exercises designed to reinforce learnings pertaining to these three vaccine-preventable diseases and their vaccinations. The components of these interventions will be designed to address specific barriers to vaccination identified by literature search and our prior work in the area of community-based vaccine education. Both arms will focus primarily on pneumococcal disease and zoster but will include limited content on influenza because participants are likely to have questions about how the flu and its vaccination differ from pneumococcal diseases and zoster. The study will be implemented in an older, predominantly African-American (AA) population, consistent with our prior work in this area.

DETAILED DESCRIPTION:
In the pharmacist-led ("PHARM") intervention group, participants will be given a 60-minute formal didactic presentation on vaccine-preventable diseases and vaccination. This presentation will be designed to address knowledge and beliefs related to zoster, pneumonia, and influenza, as well as barriers to receiving vaccination. It will be delivered by a pharmacist, will be appropriate for the participants' educational level, and will aim to establish an understanding of vaccine-preventable illnesses. The presentation will specifically discuss the following: causes, symptoms and potential complications of infections in the three diseases of interest (pneumococcal disease, zoster, and influenza); risk factors for developing the infections; incidence and prevalence of each disease of interest; modes of transmission; and disease prevention through vaccination. To improve the interactivity of the presentation, brief 30-60 second video clips excerpted from interviews with community members and physicians will be shown. Community member clips will consist of older adults from the African-American (AA) population who have experienced vaccine-preventable infections. These clips will provide culturally relevant testimony to the program audience and reinforce participant understanding of concepts introduced during didactic teaching.

In the peer-led ("PEER") intervention, peer educators will be recruited from an experienced cohort of peer educators at our senior center partner site. A pharmacist will train the peer educators about vaccine-preventable diseases over the course of two didactic sessions. Following this training, a third session will be held to train the peer educators on the script that they will deliver to participants. The script will include the key learning points to be taught by the peer educators to participants about vaccine preventable diseases and vaccination. The script will also include roleplay exercises. In the roleplay exercises, 3 scripted vaccination-related scenarios (one for each disease of interest) will be acted out by participants to illustrate scenarios participants might encounter when interacting with healthcare providers or friends/family. The skit and roleplay exercises will be practiced as needed, under the leadership of the senior center's project manager, to ensure that the peer educators are confident and consistent when delivering PEER. After completing the training, peer educators' competency on PEER program content will be assessed through a formal multiple-choice knowledge test. Each peer educator must achieve a minimum score of 80% correct over all items assessed, and 100% correct for all items deemed "core" knowledge. Once peer educator competency has been established, each peer educator will deliver PEER through a 60-minute small group session. During this session, peer educators will deliver the educational objectives through an informal discussion and will lead the group through the roleplay exercises. Participants will then be asked what key points they learned about vaccine-preventable diseases and vaccines. Finally, the peer educator will engage in a dialogue to clarify and summarize these key points.

Objectives are:

1. Compare the efficacy of PHARM vs. PEER at improving participant's knowledge regarding vaccine-preventable diseases
2. Compare the efficacy of PHARM vs. PEER at improving participants' beliefs about vaccination
3. Measure the costs of PHARM and PEER from the senior center perspective
4. Compare the percent of participants taking activation step(s) to get vaccinated following receipt of PHARM vs. PEER
5. Determine the extent to which participants are satisfied with and trust the PHARM vs. PEER interventions

Hypotheses supporting these objective are:

1. PHARM and PEER will achieve similar improvements in older adults' knowledge of vaccine preventable diseases (primary hypothesis)
2. PHARM and PEER will improved beliefs about vaccine-preventable disease
3. PEER will be a lower cost approach to educating participants in the senior center compared to PHARM
4. PHARM and PEER will result in similar rates of participants taking one or more activation step(s) to obtain vaccination
5. Participants will be highly satisfied with the PHARM and PEER interventions

ELIGIBILITY:
Inclusion Criteria:

* Age ≥50;
* Can attend a 2-hour session (though both PHARM and PEER entail 60 minutes of intervention, an additional hour is needed to allow for informed consent and data collection);
* Speak and read English at ≥4th grade level as determined by a brief reading passage;
* Cognitively intact as evidenced by an Abbreviated Mental Status Test score ≥7.

Exclusion Criteria:

* Failure to meet inclusion criteria
* Failure to give informed consent to participate in the study

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 335 (Actual)
Dates: Start 2017-10-10 (Actual); Primary Completion 2018-09-28 (Actual); Study Completion 2019-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura T Pizzi, PharmD, MPH, Principal Investigator — Rutgers University
Locations (1):
- Rutgers University, Piscataway, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
No IPD will be made available to any researchers external to this study.

REFERENCES:
- [Background] Prioli K, Schafer J, Fields Harris L, McCoy M, Barber E, Marthol-Clark M, Pizzi LT. Awareness and beliefs about pneumococcal and influenza vaccination among older African Americans: Results from a survey of community-dwelling participants at an urban senior center. Poster presented at: The 18th Annual International Meeting of the International Society for Pharmacoeconomics and Outcomes Research; May 20, 2013; New Orleans, Louisiana.
- [Background] Tomczyk S, Bennett NM, Stoecker C, Gierke R, Moore MR, Whitney CG, Hadler S, Pilishvili T; Centers for Disease Control and Prevention (CDC). Use of 13-valent pneumococcal conjugate vaccine and 23-valent pneumococcal polysaccharide vaccine among adults aged >/=65 years: recommendations of the Advisory Committee on Immunization Practices (ACIP). MMWR Morb Mortal Wkly Rep. 2014 Sep 19;63(37):822-5. PMID 25233284
- [Background] Forbes HJ, Thomas SL, Langen SM. The epidemiology and prevention of herpes zoster. Curr Derm Rep 2012;1:39-47
- [Background] Yawn BP, Saddier P, Wollan PC, St Sauver JL, Kurland MJ, Sy LS. A population-based study of the incidence and complication rates of herpes zoster before zoster vaccine introduction. Mayo Clin Proc. 2007 Nov;82(11):1341-9. doi: 10.4065/82.11.1341. PMID 17976353
- [Background] Schmader KE, Johnson GR, Saddier P, Ciarleglio M, Wang WW, Zhang JH, Chan IS, Yeh SS, Levin MJ, Harbecke RM, Oxman MN; Shingles Prevention Study Group. Effect of a zoster vaccine on herpes zoster-related interference with functional status and health-related quality-of-life measures in older adults. J Am Geriatr Soc. 2010 Sep;58(9):1634-41. doi: 10.1111/j.1532-5415.2010.03021.x. PMID 20863322
- [Background] Williams WW, Lu PJ, O'Halloran A, Bridges CB, Kim DK, Pilishvili T, Hales CM, Markowitz LE; Centers for Disease Control and Prevention (CDC). Vaccination coverage among adults, excluding influenza vaccination - United States, 2013. MMWR Morb Mortal Wkly Rep. 2015 Feb 6;64(4):95-102. PMID 25654611
- [Background] Pizzi LT, Jutkowitz E, Frick KD, Suh DC, Prioli KM, Gitlin LN. Cost-effectiveness of a community-integrated home-based depression intervention in older African Americans. J Am Geriatr Soc. 2014 Dec;62(12):2288-95. doi: 10.1111/jgs.13146. PMID 25516025
- [Background] Gitlin LN, Harris LF, McCoy MC, Chernett NL, Pizzi LT, Jutkowitz E, Hess E, Hauck WW. A home-based intervention to reduce depressive symptoms and improve quality of life in older African Americans: a randomized trial. Ann Intern Med. 2013 Aug 20;159(4):243-52. doi: 10.7326/0003-4819-159-4-201308200-00005. PMID 24026257
- [Background] Gitlin LN, Harris LF, McCoy M, Chernett NL, Jutkowitz E, Pizzi LT; Beat the Blues Team. A community-integrated home based depression intervention for older African Americans: [corrected] description of the Beat the Blues randomized trial and intervention costs. BMC Geriatr. 2012 Feb 10;12:4. doi: 10.1186/1471-2318-12-4. PMID 22325065
- [Background] Hark L, Waisbourd M, Myers JS, Henderer J, Crews JE, Saaddine JB, Molineaux J, Johnson D, Sembhi H, Stratford S, Suleiman A, Pizzi L, Spaeth GL, Katz LJ. Improving Access to Eye Care among Persons at High-Risk of Glaucoma in Philadelphia--Design and Methodology: The Philadelphia Glaucoma Detection and Treatment Project. Ophthalmic Epidemiol. 2016;23(2):122-130. doi: 10.3109/09286586.2015.1099683. Epub 2016 Mar 7. PMID 26950056
- [Background] Waisbourd M, Shafa A, Delvadia R, Sembhi H, Molineaux J, Henderer J, Pizzi LT, Myers JS, Hark LA, Katz LJ. Bilateral Same-day Laser Peripheral Iridotomy in the Philadelphia Glaucoma Detection and Treatment Project. J Glaucoma. 2016 Oct;25(10):e821-e825. doi: 10.1097/IJG.0000000000000409. PMID 26950579
- [Background] Alcusky MJ, Cannon-Dang E, Steele D, Schafer JJ, DeSimone Jr. JA, Pizzi LT. Cost of a pharmacist-led pneumonia education and immunization program for older Philadelphians. Poster presentation at the ISPOR 20th Annual International Meeting, May 16-20 2015 Philadelphia, PA.
- [Background] Schafer JJ, Steele D, Marthol MM, Harris LF, Pizzi LT. Knowledge gaps about pneumonia in older adults: results from the pharmacists' pneumonia prevention project. Poster presentation at the ISPOR 20th Annual International Meeting, May 16-20, 2015 Philadelphia, PA.
- [Background] Pizzi LT, Steele D, Sembhi H, Hark L, Waisbourd M, Katz LJ. Cost analysis of the Philadelphia glaucoma community detection and treatment project. Poster presentation at the ISPOR 20th Annual International Meeting, May 16-20, 2015 Philadelphia, PA.
- [Background] Luque JS, Ross L, Gwede CK. Qualitative systematic review of barber-administered health education, promotion, screening and outreach programs in African-American communities. J Community Health. 2014 Feb;39(1):181-90. doi: 10.1007/s10900-013-9744-3. PMID 23913106
- [Background] Linnan LA, D'Angelo H, Harrington CB. A literature synthesis of health promotion research in salons and barbershops. Am J Prev Med. 2014 Jul;47(1):77-85. doi: 10.1016/j.amepre.2014.02.007. Epub 2014 Apr 24. PMID 24768037
- [Background] Schulman-Green D, Jaser S, Martin F, Alonzo A, Grey M, McCorkle R, Redeker NS, Reynolds N, Whittemore R. Processes of self-management in chronic illness. J Nurs Scholarsh. 2012 Jun;44(2):136-44. doi: 10.1111/j.1547-5069.2012.01444.x. Epub 2012 May 2. PMID 22551013
- [Background] Swendeman D, Ingram BL, Rotheram-Borus MJ. Common elements in self-management of HIV and other chronic illnesses: an integrative framework. AIDS Care. 2009 Oct;21(10):1321-34. doi: 10.1080/09540120902803158. PMID 20024709
- [Background] Kennedy DT, Small RE. Development and implementation of a smoking cessation clinic in community pharmacy practice. J Am Pharm Assoc (Wash). 2002 Jan-Feb;42(1):83-92. doi: 10.1331/108658002763538116. PMID 11833523
- [Background] American Pharmacists Association; National Association of Chain Drug Stores Foundation. Medication therapy management in pharmacy practice: core elements of an MTM service model (version 2.0). J Am Pharm Assoc (2003). 2008 May-Jun;48(3):341-53. doi: 10.1331/JAPhA.2008.08514. PMID 18595820
- [Background] Centers for Disease Control and Prevention (CDC); Advisory Committee on Immunization Practices. Updated recommendations for prevention of invasive pneumococcal disease among adults using the 23-valent pneumococcal polysaccharide vaccine (PPSV23). MMWR Morb Mortal Wkly Rep. 2010 Sep 3;59(34):1102-6. PMID 20814406
- [Background] Schneeberg A, Bettinger JA, McNeil S, Ward BJ, Dionne M, Cooper C, Coleman B, Loeb M, Rubinstein E, McElhaney J, Scheifele DW, Halperin SA. Knowledge, attitudes, beliefs and behaviours of older adults about pneumococcal immunization, a Public Health Agency of Canada/Canadian Institutes of Health Research Influenza Research Network (PCIRN) investigation. BMC Public Health. 2014 May 12;14:442. doi: 10.1186/1471-2458-14-442. PMID 24884433
- [Background] Lu PJ, Euler GL, Jumaan AO, Harpaz R. Herpes zoster vaccination among adults aged 60 years or older in the United States, 2007: uptake of the first new vaccine to target seniors. Vaccine. 2009 Feb 5;27(6):882-7. doi: 10.1016/j.vaccine.2008.11.077. Epub 2008 Dec 9. PMID 19071175
- [Background] Hurley LP, Harpaz R, Daley MF, Crane LA, Beaty BL, Barrow J, Babbel C, Marin M, Steiner JF, Davidson A, Dickinson LM, Kempe A. National survey of primary care physicians regarding herpes zoster and the herpes zoster vaccine. J Infect Dis. 2008 Mar 1;197 Suppl 2:S216-23. doi: 10.1086/522153. PMID 18419400
- [Background] Hurley LP, Lindley MC, Harpaz R, Stokley S, Daley MF, Crane LA, Dong F, Beaty BL, Tan L, Babbel C, Dickinson LM, Kempe A. Barriers to the use of herpes zoster vaccine. Ann Intern Med. 2010 May 4;152(9):555-60. doi: 10.7326/0003-4819-152-9-201005040-00005. PMID 20439573
- [Background] Zimmerman RK, Santibanez TA, Fine MJ, Janosky JE, Nowalk MP, Bardella IJ, Raymund M, Wilson SA. Barriers and facilitators of pneumococcal vaccination among the elderly. Vaccine. 2003 Mar 28;21(13-14):1510-7. doi: 10.1016/s0264-410x(02)00698-9. PMID 12615448
- [Background] Harris LM, Chin NP, Fiscella K, Humiston S. Barrier to pneumococcal and influenza vaccinations in Black elderly communities: mistrust. J Natl Med Assoc. 2006 Oct;98(10):1678-84. PMID 17052061
- [Background] Nowalk MP, Zimmerman RK, Shen S, Jewell IK, Raymund M. Barriers to pneumococcal and influenza vaccination in older community-dwelling adults (2000-2001). J Am Geriatr Soc. 2004 Jan;52(1):25-30. doi: 10.1111/j.1532-5415.2004.52006.x. PMID 14687311
- [Background] Hoffmann S, Caro FG, Gottlieb AS, Kesternich I, Winter JK. Contributions of Second Opinions, Outcome Forecasts, and Testimonials to Patient Decisions about Knee Replacement Surgery. Med Decis Making. 2014 Jul;34(5):603-14. doi: 10.1177/0272989X14527796. Epub 2014 Apr 16. PMID 24739534
- [Background] Ubel PA, Jepson C, Baron J. The inclusion of patient testimonials in decision aids: effects on treatment choices. Med Decis Making. 2001 Jan-Feb;21(1):60-8. doi: 10.1177/0272989X0102100108. PMID 11206948
- [Background] Singleton JA, Santibanez TA, Wortley PM. Influenza and pneumococcal vaccination of adults aged > or = 65: racial/ethnic differences. Am J Prev Med. 2005 Dec;29(5):412-20. doi: 10.1016/j.amepre.2005.08.012. PMID 16376704
- [Background] Mieczkowski TA, Wilson SA. Adult pneumococcal vaccination: a review of physician and patient barriers. Vaccine. 2002 Jan 31;20(9-10):1383-92. doi: 10.1016/s0264-410x(01)00463-7. PMID 11818157
- [Background] Jones LG, Zhang Y, Ahmed MI, Ekundayo OJ, Akhter S, Sawyer P, Aban I, Sims RV, Ahmed A. Understanding the reasons for the underuse of pneumococcal vaccination by community-dwelling older African Americans. J Am Geriatr Soc. 2010 Dec;58(12):2323-8. doi: 10.1111/j.1532-5415.2010.03181.x. PMID 21143440
- [Background] Santibanez TA, Nowalk MP, Zimmerman RK, Jewell IK, Bardella IJ, Wilson SA, Terry MA. Knowledge and beliefs about influenza, pneumococcal disease, and immunizations among older people. J Am Geriatr Soc. 2002 Oct;50(10):1711-6. doi: 10.1046/j.1532-5415.2002.50466.x. PMID 12366627
- [Derived] Prioli KM, Akincigil A, Namvar T, Mitchell-Williams J, Schafer JJ, Cunningham RC, Fields-Harris L, McCoy M, Vertsman R, Guesnier A, Pizzi LT. Addressing racial inequality and its effects on vaccination rate: A trial comparing a pharmacist and peer educational program (MOTIVATE) in diverse older adults. J Manag Care Spec Pharm. 2023 Aug;29(8):970-980. doi: 10.18553/jmcp.2023.29.8.970. PMID 37523315
- See also: Immunization Action Coalition. Pneumococcal Polysaccharide Vaccination Pocket Guide. — http://www.immunize.org/catg.d/p4213.pdf

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pharmacist-led Intervention (PHARM) | Peer-led Intervention (PEER)
Started | 175 | 160
Met Inclusion Criteria | 150 | 144
Submitted Survey Data | 147 | 140
Completed | 147 | 140
Not Completed | 28 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pharmacist-led Intervention (PHARM) | Peer-led Intervention (PEER) | Total
Number analyzed (Participants) | 147 | 140 | 287
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.2 (9.17) | 73.9 (8.67) | 74.5 (8.94)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 118 | 113 | 231
  Male | 25 | 26 | 51
  I prefer not to answer / No response | 4 | 1 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 68 | 115 | 183
  White | 61 | 16 | 77
  Asian | 7 | 1 | 8
  Latino | 0 | 3 | 3
  Other | 5 | 2 | 7
  I don't know / Not sure | 1 | 0 | 1
  I prefer not to answer / No response | 5 | 3 | 8
Region of Enrollment [Number; unit: participants]
  United States | 147 | 140 | 287
Highest degree of education achieved [Count of Participants; unit: Participants]
  High school graduate or GED | 61 | 55 | 116
  Some college or vocational school | 35 | 41 | 76
  College graduate | 30 | 32 | 62
  I prefer not to answer / No response | 21 | 12 | 33
Marital Status [Count of Participants; unit: Participants]
  Never married | 26 | 22 | 48
  Married or living as married | 21 | 25 | 46
  Widowed, not currently married | 62 | 49 | 111
  Divorced, not currently married | 25 | 29 | 54
  Separated | 6 | 10 | 16
  I don't know / Not sure | 1 | 0 | 1
  I prefer not to answer / No response | 6 | 5 | 11
Difficulty paying for basic necessities [Count of Participants; unit: Participants]
  Not difficult at all | 57 | 61 | 118
  Not very difficult | 33 | 31 | 64
  Somewhat difficult | 31 | 29 | 60
  Very difficult | 8 | 11 | 19
  I don't know / not sure | 3 | 2 | 5
  I prefer not to answer / No response | 15 | 6 | 21
Baseline Knowledge Scores [Mean (Standard Deviation); unit: Scores on a scale] — Knowledge and awareness about the target vaccine-preventable diseases was assessed at baseline using the Knowledge Instrument, a 3-section, 22-item instrument categorical response instrument. Scores consist of number of correct responses to the questions on the knowledge instrument; a higher score indicates better performance. Four scores are possible: 3 disease-specific subscores (1 each for pneumonia, influenza, and zoster) and 1 total score (equaling the sum of the 3 disease-specific subscores). Possible score ranges are as follows: pneumonia 0-7; influenza 0-7; zoster 0-8; total 0-22.
  Scores on a scale
    Total Knowledge Score (number correct out of 22) | 11.6 (4.80) | 12.0 (4.82) | 11.8 (4.81)
    Zoster Knowledge Score (number correct out of 8) | 3.8 (1.99) | 3.9 (1.96) | 3.85 (1.97)
    Pneumonia Knowledge Score (# correct out of 7) | 3.1 (2.03) | 3.4 (2.05) | 3.3 (2.04)
    Influenza Knowledge Score (# correct out of 7) | 4.8 (1.69) | 4.8 (1.63) | 4.8 (1.66)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Knowledge and Awareness About Vaccine-Preventable Diseases
Description: Knowledge and awareness about the target vaccine-preventable diseases was assessed at each timepoint using the VEPSC Knowledge Instrument, a 3-section, 22-item instrument categorical response instrument. Scores consist of number of correct responses to the questions on the knowledge instrument, thus a higher score indicates better performance. Four scores are possible: three disease-specific subscores (one each for pneumonia, influenza, and zoster) and one total score (equaling the sum of the three disease-specific subscores). Possible score ranges are as follows: pneumonia 0-7; influenza 0-7; zoster 0-8; total 0-22. For each score type, pairwise score differences were calculated between all 3 timepoints (baseline, post-test, and one-month follow-up). Positive values indicate increased knowledge among participants; negative values indicate decreased knowledge.
Time Frame: Measured at baseline (BL), immediately post-intervention (PT), and 1 month follow-up (1M)
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Pharmacist-led Intervention (PHARM) | Peer-led Intervention (PEER)
Number analyzed (Participants) | 147 | 140
Scores on a scale
  Baseline to Post Test score change - Total | 3.5 (4.03) | 4.9 (4.25)
  Baseline to Post Test score change - Zoster | 1.3 (1.85) | 1.8 (1.86)
  Baseline to Post Test score change - Pneumonia | 1.5 (1.89) | 1.9 (1.97)
  Baseline to Post Test change - Influenza | 0.5 (1.38) | 1.1 (1.58)
  Baseline to 1 month follow up change - Total | 3.4 (4.22) | 4.3 (4.82)
  Baseline to 1 month follow up change - Zoster | 1.3 (1.97) | 1.5 (2.04)
  Baseline to 1 month follow up change - Pneumonia | 1.5 (1.83) | 1.5 (2.22)
  Baseline to 1 month follow up change - Influenza | 0.5 (1.49) | 1.2 (1.83)
  Post test to 1 month follow up change - Total | -0.15 (2.26) | -0.6 (3.51)
  Post test to 1 month follow up change - Zoster | -0.03 (0.90) | -0.2 (1.46)
  Post test to 1 month follow up change - Pneumonia | -0.09 (1.94) | -0.4 (1.76)
  Post test to 1 month follow up change - Influenza | -0.03 (0.89) | 0.04 (0.6973)
Statistical Analysis 1: Comparison: Pharmacist-led Intervention (PHARM) vs Peer-led Intervention (PEER); Testing total knowledge score change between groups from baseline to post intervention; Test type: Equivalence — Two-sided Wilcoxon Rank-Sum test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons); p = 0.0081, Wilcoxon (Mann-Whitney) — Two-sided Wilcoxon Rank-Sum test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons)
Statistical Analysis 2: Comparison: Pharmacist-led Intervention (PHARM) vs Peer-led Intervention (PEER); Testing zoster knowledge score change between groups from baseline to post intervention; Test type: Equivalence — Two-sided Wilcoxon Rank-Sum test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons); p = 0.0243, Wilcoxon (Mann-Whitney) — Two-sided Wilcoxon Rank-Sum test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons)
Statistical Analysis 3: Comparison: Pharmacist-led Intervention (PHARM) vs Peer-led Intervention (PEER); Testing pneumonia knowledge score change between groups from baseline to post intervention; Test type: Equivalence — Two-sided Wilcoxon Rank-Sum test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons); p = 0.0710, Wilcoxon (Mann-Whitney) — Two-sided Wilcoxon Rank-Sum test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons)
Statistical Analysis 4: Comparison: Pharmacist-led Intervention (PHARM) vs Peer-led Intervention (PEER); Testing influenza knowledge score change between groups from baseline to post intervention; Test type: Equivalence — Two-sided Wilcoxon Rank-Sum test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons); p = 0.0008, Wilcoxon (Mann-Whitney) — Two-sided Wilcoxon Rank-Sum test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons)
Statistical Analysis 5: Comparison: Pharmacist-led Intervention (PHARM) vs Peer-led Intervention (PEER); Testing total knowledge score change between groups from baseline to one-month follow-up; Test type: Equivalence — Two-sided Wilcoxon Rank-Sum test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons); p = 0.1094, Wilcoxon (Mann-Whitney) — Two-sided Wilcoxon Rank-Sum test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons)
Statistical Analysis 6: Comparison: Pharmacist-led Intervention (PHARM) vs Peer-led Intervention (PEER); Testing zoster knowledge score change between groups from baseline to one-month follow-up; Test type: Equivalence — Two-sided Wilcoxon Rank-Sum test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons); p = 0.2029, Wilcoxon (Mann-Whitney) — Two-sided Wilcoxon Rank-Sum test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons)
Statistical Analysis 7: Comparison: Pharmacist-led Intervention (PHARM) vs Peer-led Intervention (PEER); Testing pneumonia knowledge score change between groups from baseline to one-month follow-up; Test type: Equivalence — Two-sided Wilcoxon Rank-Sum test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons); p = 0.8599, Wilcoxon (Mann-Whitney) — Two-sided Wilcoxon Rank-Sum test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons)
Statistical Analysis 8: Comparison: Pharmacist-led Intervention (PHARM) vs Peer-led Intervention (PEER); Testing influenza knowledge score change between groups from baseline to one-month follow-up; Test type: Equivalence — Two-sided Wilcoxon Rank-Sum test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons); p = 0.0007, Wilcoxon (Mann-Whitney) — Two-sided Wilcoxon Rank-Sum test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons)
Statistical Analysis 9: Comparison: Pharmacist-led Intervention (PHARM) vs Peer-led Intervention (PEER); Testing total knowledge score change between groups from post-intervention to one-month follow-up; Test type: Equivalence — Two-sided Wilcoxon Rank-Sum test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons); p = 0.0246, Wilcoxon (Mann-Whitney) — Two-sided Wilcoxon Rank-Sum test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons)
Statistical Analysis 10: Comparison: Pharmacist-led Intervention (PHARM) vs Peer-led Intervention (PEER); Testing zoster knowledge score change between groups from post-intervention to one-month follow-up; Test type: Equivalence — Two-sided Wilcoxon Rank-Sum test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons); p = 0.0780, Wilcoxon (Mann-Whitney) — Two-sided Wilcoxon Rank-Sum test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons)
Statistical Analysis 11: Comparison: Pharmacist-led Intervention (PHARM) vs Peer-led Intervention (PEER); Testing pneumonia knowledge score change between groups from post-intervention to one-month follow-up; Test type: Equivalence — Two-sided Wilcoxon Rank-Sum test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons); p = 0.0167, Wilcoxon (Mann-Whitney) — Two-sided Wilcoxon Rank-Sum test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons)
Statistical Analysis 12: Comparison: Pharmacist-led Intervention (PHARM) vs Peer-led Intervention (PEER); Testing influenza knowledge score change between groups from post-intervention to one-month follow-up; Test type: Equivalence — Two-sided Wilcoxon Rank-Sum test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons); p = 0.9417, Wilcoxon (Mann-Whitney) — Two-sided Wilcoxon Rank-Sum test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons)

2. Secondary Outcome: Within-Group Changes in Beliefs About Vaccine-Preventable Diseases and Vaccines
Description: Beliefs about vaccine-preventable diseases and vaccination were assessed via agreement with 5 statements scored on a 4-point Likert scale (1-Completely disagree, 2-Somewhat disagree, 3-Somewhat agree, 4-Completely agree) at each timepoint. The changes in beliefs between baseline, post-intervention, and the one-month follow-up were assessed in both PHARM and PEER groups. Pairwise Wilcoxon Signed-Rank tests were run comparing within-group changes in beliefs across timepoints and applying the Bonferroni correction (α=0.05/3=0.0167).
Time Frame: Measured at baseline (BL), immediately post-intervention (PT), and 1 month follow-up (1M)
Measure: Count of Participants; unit: Participants
Arm/Group | Pharmacist-led Intervention (PHARM) | Peer-led Intervention (PEER)
Number analyzed (Participants) | 147 | 140
Participants
  Vaccinations are important for health (BL to PT): Strongly decreased agreement (3-point decrease) | 1 | 0
  Vaccinations are important for health (BL to PT): Somewhat decreased agreement (2-point decrease) | 0 | 0
  Vaccinations are important for health (BL to PT): Slightly decreased agreement (1-point decrease) | 3 | 1
  Vaccinations are important for health (BL to PT): No change in agreement | 108 | 97
  Vaccinations are important for health (BL to PT): Slightly improved agreement (1-point increase) | 19 | 27
  Vaccinations are important for health (BL to PT): Somewhat improved agreement (2-point increase) | 2 | 5
  Vaccinations are important for health (BL to PT): Strongly improved agreement (3-point increase) | 0 | 2
  Vaccinations are important for health (BL to PT): No response | 14 | 8
  Vaccinations are important for health (BL to 1M): Strongly decreased agreement (3-point decrease) | 1 | 1
  Vaccinations are important for health (BL to 1M): Somewhat decreased agreement (2-point decrease) | 0 | 0
  Vaccinations are important for health (BL to 1M): Slightly decreased agreement (1-point decrease) | 4 | 2
  Vaccinations are important for health (BL to 1M): No change in agreement | 107 | 94
  Vaccinations are important for health (BL to 1M): Slightly improved agreement (1-point increase) | 19 | 28
  Vaccinations are important for health (BL to 1M): Somewhat improved agreement (2-point increase) | 2 | 5
  Vaccinations are important for health (BL to 1M): Strongly improved agreement (3-point increase) | 0 | 2
  Vaccinations are important for health (BL to 1M): No response | 14 | 8
  Vaccinations are important for health (PT to 1M): Strongly decreased agreement (3-point decrease) | 0 | 2
  Vaccinations are important for health (PT to 1M): Somewhat decreased agreement (2-point decrease) | 0 | 1
  Vaccinations are important for health (PT to 1M): Slightly decreased agreement (1-point decrease) | 3 | 6
  Vaccinations are important for health (PT to 1M): No change in agreement | 139 | 122
  Vaccinations are important for health (PT to 1M): Slightly improved agreement (1-point increase) | 2 | 8
  Vaccinations are important for health (PT to 1M): Somewhat improved agreement (2-point increase) | 0 | 1
  Vaccinations are important for health (PT to 1M): Strongly improved agreement (3-point increase) | 0 | 0
  Vaccinations are important for health (PT to 1M): No response | 3 | 0
  Vaccines are harmful to health (BL to PT): Strongly decreased agreement (3-point decrease) | 3 | 7
  Vaccines are harmful to health (BL to PT): Somewhat decreased agreement (2-point decrease) | 7 | 13
  Vaccines are harmful to health (BL to PT): Slightly decreased agreement (1-point decrease) | 9 | 12
  Vaccines are harmful to health (BL to PT): No change in agreement | 79 | 53
  Vaccines are harmful to health (BL to PT): Slightly improved agreement (1-point increase) | 4 | 7
  Vaccines are harmful to health (BL to PT): Somewhat improved agreement (2-point increase) | 3 | 1
  Vaccines are harmful to health (BL to PT): Strongly improved agreement (3-point increase) | 2 | 0
  Vaccines are harmful to health (BL to PT): No response | 40 | 47
  Vaccines are harmful to health (BL to 1M): Strongly decreased agreement (3-point decrease) | 3 | 6
  Vaccines are harmful to health (BL to 1M): Somewhat decreased agreement (2-point decrease) | 7 | 13
  Vaccines are harmful to health (BL to 1M): Slightly decreased agreement (1-point decrease) | 12 | 21
  Vaccines are harmful to health (BL to 1M): No change in agreement | 70 | 38
  Vaccines are harmful to health (BL to 1M): Slightly improved agreement (1-point increase) | 6 | 11
  Vaccines are harmful to health (BL to 1M): Somewhat improved agreement (2-point increase) | 7 | 3
  Vaccines are harmful to health (BL to 1M): Strongly improved agreement (3-point increase) | 2 | 1
  Vaccines are harmful to health (BL to 1M): No response | 40 | 47
  Vaccines are harmful to health (PT to 1M): Strongly decreased agreement (3-point decrease) | 2 | 3
  Vaccines are harmful to health (PT to 1M): Somewhat decreased agreement (2-point decrease) | 2 | 5
  Vaccines are harmful to health (PT to 1M): Slightly decreased agreement (1-point decrease) | 6 | 10
  Vaccines are harmful to health (PT to 1M): No change in agreement | 111 | 83
  Vaccines are harmful to health (PT to 1M): Slightly improved agreement (1-point increase) | 9 | 15
  Vaccines are harmful to health (PT to 1M): Somewhat improved agreement (2-point increase) | 6 | 8
  Vaccines are harmful to health (PT to 1M): Strongly improved agreement (3-point increase) | 1 | 2
  Vaccines are harmful to health (PT to 1M): No response | 10 | 14
  Trust in doctors as vaccine info source (BL to PT): Strongly decreased agreement (3-point decrease) | 0 | 1
  Trust in doctors as vaccine info source (BL to PT): Somewhat decreased agreement (2-point decrease) | 0 | 2
  Trust in doctors as vaccine info source (BL to PT): Slightly decreased agreement (1-point decrease) | 6 | 5
  Trust in doctors as vaccine info source (BL to PT): No change in agreement | 117 | 102
  Trust in doctors as vaccine info source (BL to PT): Slightly improved agreement (1-point increase) | 10 | 19
  Trust in doctors as vaccine info source (BL to PT): Somewhat improved agreement (2-point increase) | 2 | 3
  Trust in doctors as vaccine info source (BL to PT): Strongly improved agreement (3-point increase) | 0 | 0
  Trust in doctors as vaccine info source (BL to PT): No response | 12 | 8
  Trust in doctors as vaccine info source (BL to 1M): Strongly decreased agreement (3-point decrease) | 1 | 1
  Trust in doctors as vaccine info source (BL to 1M): Somewhat decreased agreement (2-point decrease) | 0 | 2
  Trust in doctors as vaccine info source (BL to 1M): Slightly decreased agreement (1-point decrease) | 10 | 5
  Trust in doctors as vaccine info source (BL to 1M): No change in agreement | 112 | 98
  Trust in doctors as vaccine info source (BL to 1M): Slightly improved agreement (1-point increase) | 10 | 20
  Trust in doctors as vaccine info source (BL to 1M): Somewhat improved agreement (2-point increase) | 2 | 6
  Trust in doctors as vaccine info source (BL to 1M): Strongly improved agreement (3-point increase) | 0 | 0
  Trust in doctors as vaccine info source (BL to 1M): No response | 12 | 8
  Trust in doctors as vaccine info source (PT to 1M): Strongly decreased agreement (3-point decrease) | 1 | 3
  Trust in doctors as vaccine info source (PT to 1M): Somewhat decreased agreement (2-point decrease) | 1 | 0
  Trust in doctors as vaccine info source (PT to 1M): Slightly decreased agreement (1-point decrease) | 4 | 6
  Trust in doctors as vaccine info source (PT to 1M): No change in agreement | 137 | 115
  Trust in doctors as vaccine info source (PT to 1M): Slightly improved agreement (1-point increase) | 2 | 10
  Trust in doctors as vaccine info source (PT to 1M): Somewhat improved agreement (2-point increase) | 0 | 4
  Trust in doctors as vaccine info source (PT to 1M): Strongly improved agreement (3-point increase) | 0 | 1
  Trust in doctors as vaccine info source (PT to 1M): No response | 2 | 1
  Trust in pharmacists for vaccine info (BL to PT): Strongly decreased agreement (3-point decrease) | 2 | 0
  Trust in pharmacists for vaccine info (BL to PT): Somewhat decreased agreement (2-point decrease) | 1 | 1
  Trust in pharmacists for vaccine info (BL to PT): Slightly decreased agreement (1-point decrease) | 4 | 11
  Trust in pharmacists for vaccine info (BL to PT): No change in agreement | 112 | 96
  Trust in pharmacists for vaccine info (BL to PT): Slightly improved agreement (1-point increase) | 12 | 21
  Trust in pharmacists for vaccine info (BL to PT): Somewhat improved agreement (2-point increase) | 0 | 3
  Trust in pharmacists for vaccine info (BL to PT): Strongly improved agreement (3-point increase) | 1 | 1
  Trust in pharmacists for vaccine info (BL to PT): No response | 15 | 7
  Trust in pharmacists for vaccine info (BL to 1M): Strongly decreased agreement (3-point decrease) | 3 | 1
  Trust in pharmacists for vaccine info (BL to 1M): Somewhat decreased agreement (2-point decrease) | 3 | 2
  Trust in pharmacists for vaccine info (BL to 1M): Slightly decreased agreement (1-point decrease) | 13 | 14
  Trust in pharmacists for vaccine info (BL to 1M): No change in agreement | 99 | 84
  Trust in pharmacists for vaccine info (BL to 1M): Slightly improved agreement (1-point increase) | 12 | 28
  Trust in pharmacists for vaccine info (BL to 1M): Somewhat improved agreement (2-point increase) | 0 | 4
  Trust in pharmacists for vaccine info (BL to 1M): Strongly improved agreement (3-point increase) | 2 | 0
  Trust in pharmacists for vaccine info (BL to 1M): No response | 15 | 7
  Trust in pharmacists for vaccine info (PT to 1M): Strongly decreased agreement (3-point decrease) | 1 | 4
  Trust in pharmacists for vaccine info (PT to 1M): Somewhat decreased agreement (2-point decrease) | 4 | 2
  Trust in pharmacists for vaccine info (PT to 1M): Slightly decreased agreement (1-point decrease) | 7 | 13
  Trust in pharmacists for vaccine info (PT to 1M): No change in agreement | 129 | 98
  Trust in pharmacists for vaccine info (PT to 1M): Slightly improved agreement (1-point increase) | 3 | 19
  Trust in pharmacists for vaccine info (PT to 1M): Somewhat improved agreement (2-point increase) | 0 | 1
  Trust in pharmacists for vaccine info (PT to 1M): Strongly improved agreement (3-point increase) | 1 | 1
  Trust in pharmacists for vaccine info (PT to 1M): No response | 2 | 2
  Trust in peer educators for vaccine info(BL to PT): Strongly decreased agreement (3-point decrease) | 2 | 0
  Trust in peer educators for vaccine info(BL to PT): Somewhat decreased agreement (2-point decrease) | 5 | 5
  Trust in peer educators for vaccine info(BL to PT): Slightly decreased agreement (1-point decrease) | 7 | 12
  Trust in peer educators for vaccine info(BL to PT): No change in agreement | 86 | 77
  Trust in peer educators for vaccine info(BL to PT): Slightly improved agreement (1-point increase) | 19 | 27
  Trust in peer educators for vaccine info(BL to PT): Somewhat improved agreement (2-point increase) | 2 | 3
  Trust in peer educators for vaccine info(BL to PT): Strongly improved agreement (3-point increase) | 3 | 0
  Trust in peer educators for vaccine info(BL to PT): No response | 23 | 16
  Trust in peer educators for vaccine info(BL to 1M): Strongly decreased agreement (3-point decrease) | 0 | 3
  Trust in peer educators for vaccine info(BL to 1M): Somewhat decreased agreement (2-point decrease) | 11 | 5
  Trust in peer educators for vaccine info(BL to 1M): Slightly decreased agreement (1-point decrease) | 12 | 11
  Trust in peer educators for vaccine info(BL to 1M): No change in agreement | 74 | 55
  Trust in peer educators for vaccine info(BL to 1M): Slightly improved agreement (1-point increase) | 19 | 37
  Trust in peer educators for vaccine info(BL to 1M): Somewhat improved agreement (2-point increase) | 4 | 7
  Trust in peer educators for vaccine info(BL to 1M): Strongly improved agreement (3-point increase) | 4 | 6
  Trust in peer educators for vaccine info(BL to 1M): No response | 23 | 16
  Trust in peer educators for vaccine info(PT to 1M): Strongly decreased agreement (3-point decrease) | 2 | 4
  Trust in peer educators for vaccine info(PT to 1M): Somewhat decreased agreement (2-point decrease) | 7 | 9
  Trust in peer educators for vaccine info(PT to 1M): Slightly decreased agreement (1-point decrease) | 7 | 10
  Trust in peer educators for vaccine info(PT to 1M): No change in agreement | 114 | 73
  Trust in peer educators for vaccine info(PT to 1M): Slightly improved agreement (1-point increase) | 4 | 19
  Trust in peer educators for vaccine info(PT to 1M): Somewhat improved agreement (2-point increase) | 2 | 9
  Trust in peer educators for vaccine info(PT to 1M): Strongly improved agreement (3-point increase) | 5 | 9
  Trust in peer educators for vaccine info(PT to 1M): No response | 6 | 7
Statistical Analysis 1: Comparison: Pharmacist-led Intervention (PHARM); Testing within-group changes in beliefs for the statement "Getting vaccinations is important to my health" from baseline to post-intervention; Test type: Equivalence — Wilcoxon Signed-Rank test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons); p = 0.0011, Sign test — Wilcoxon Signed-Rank test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons)
Statistical Analysis 2: Comparison: Peer-led Intervention (PEER); [analysis description as in outcome 2, analysis 1]; Test type: Equivalence — Wilcoxon Signed-Rank test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons); p < 0.0001, Sign test — Wilcoxon Signed-Rank test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons)
Statistical Analysis 3: Comparison: Pharmacist-led Intervention (PHARM); Testing within-group changes in beliefs for the statement "Getting vaccinations is important to my health" from baseline to one-month follow-up; Test type: Equivalence — Wilcoxon Signed-Rank test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons); p = 0.0028, Sign test — Wilcoxon Signed-Rank test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons)
Statistical Analysis 4: Comparison: Peer-led Intervention (PEER); [analysis description as in outcome 2, analysis 3]; Test type: Equivalence — Wilcoxon Signed-Rank test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons); p < 0.0001, Sign test — Wilcoxon Signed-Rank test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons)
Statistical Analysis 5: Comparison: Pharmacist-led Intervention (PHARM); Testing within-group changes in beliefs for the statement "Getting vaccinations is important to my health" from post-intervention to one-month follow-up; Test type: Equivalence — Wilcoxon Signed-Rank test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons); p = 1.0, Sign test — Wilcoxon Signed-Rank test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons)
Statistical Analysis 6: Comparison: Peer-led Intervention (PEER); [analysis description as in outcome 2, analysis 5]; Test type: Equivalence — Wilcoxon Signed-Rank test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons); p = 0.6430, Sign test — Wilcoxon Signed-Rank test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons)
Statistical Analysis 7: Comparison: Pharmacist-led Intervention (PHARM); Testing within-group changes in beliefs for the statement "Getting vaccinations can be harmful to my health" from baseline to post-intervention; Test type: Equivalence — Wilcoxon Signed-Rank test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons); p = 0.1193, Sign test — Wilcoxon Signed-Rank test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons)
Statistical Analysis 8: Comparison: Peer-led Intervention (PEER); [analysis description as in outcome 2, analysis 7]; Test type: Equivalence — Wilcoxon Signed-Rank test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons); p < 0.0001, Sign test — Wilcoxon Signed-Rank test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons)
Statistical Analysis 9: Comparison: Pharmacist-led Intervention (PHARM); Testing within-group changes in beliefs for the statement "Getting vaccinations can be harmful to my health" from baseline to one-month follow-up; Test type: Equivalence — Wilcoxon Signed-Rank test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons); p = 0.4861, Sign test — Wilcoxon Signed-Rank test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons)
Statistical Analysis 10: Comparison: Peer-led Intervention (PEER); [analysis description as in outcome 2, analysis 9]; Test type: Equivalence — Wilcoxon Signed-Rank test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons); p = 0.0002, Sign test — Wilcoxon Signed-Rank test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons)
Statistical Analysis 11: Comparison: Pharmacist-led Intervention (PHARM); Testing within-group changes in beliefs for the statement "Getting vaccinations can be harmful to my health" from post-intervention to one-month follow-up; Test type: Equivalence — Wilcoxon Signed-Rank test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons); p = 0.3247, Sign test — Wilcoxon Signed-Rank test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons)
Statistical Analysis 12: Comparison: Peer-led Intervention (PEER); [analysis description as in outcome 2, analysis 11]; Test type: Equivalence — Wilcoxon Signed-Rank test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons); p = 0.4627, Sign test — Wilcoxon Signed-Rank test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons)
Statistical Analysis 13: Comparison: Pharmacist-led Intervention (PHARM); Testing within-group changes in beliefs for the statement "I trust my doctor to give me information about vaccines and the diseases they prevent" from baseline to post-intervention; Test type: Equivalence — Wilcoxon Signed-Rank test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons); p = 0.1244, Sign test — Wilcoxon Signed-Rank test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons)
Statistical Analysis 14: Comparison: Peer-led Intervention (PEER); [analysis description as in outcome 2, analysis 13]; Test type: Equivalence — Wilcoxon Signed-Rank test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons); p = 0.0575, Sign test — Wilcoxon Signed-Rank test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons)
Statistical Analysis 15: Comparison: Pharmacist-led Intervention (PHARM); Testing within-group changes in beliefs for the statement "I trust my doctor to give me information about vaccines and the diseases they prevent" from baseline to one-month follow-up; Test type: Equivalence — Wilcoxon Signed-Rank test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons); p = 0.7489, Sign test — Wilcoxon Signed-Rank test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons)
Statistical Analysis 16: Comparison: Peer-led Intervention (PEER); [analysis description as in outcome 2, analysis 15]; Test type: Equivalence — Wilcoxon Signed-Rank test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons); p = 0.0098, Sign test — Wilcoxon Signed-Rank test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons)
Statistical Analysis 17: Comparison: Pharmacist-led Intervention (PHARM); Testing within-group changes in beliefs for the statement "I trust my doctor to give me information about vaccines and the diseases they prevent" from post-intervention to one-month follow-up; Test type: Equivalence — Wilcoxon Signed-Rank test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons); p = 0.1797, Sign test — Wilcoxon Signed-Rank test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons)
Statistical Analysis 18: Comparison: Peer-led Intervention (PEER); [analysis description as in outcome 2, analysis 17]; Test type: Equivalence — Wilcoxon Signed-Rank test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons); p = 0.3613, Sign test — Wilcoxon Signed-Rank test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons)
Statistical Analysis 19: Comparison: Pharmacist-led Intervention (PHARM); Testing within-group changes in beliefs for the statement "I trust my pharmacist to give me information about vaccines and the diseases they prevent" from baseline to post-intervention; Test type: Equivalence — Wilcoxon Signed-Rank test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons); p = 0.5972, Sign test — Wilcoxon Signed-Rank test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons)
Statistical Analysis 20: Comparison: Peer-led Intervention (PEER); [analysis description as in outcome 2, analysis 19]; Test type: Equivalence — Wilcoxon Signed-Rank test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons); p = 0.0240, Sign test — Wilcoxon Signed-Rank test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons)
Statistical Analysis 21: Comparison: Pharmacist-led Intervention (PHARM); Testing within-group changes in beliefs for the statement "I trust my pharmacist to give me information about vaccines and the diseases they prevent" from baseline to one-month follow-up; Test type: Equivalence — Wilcoxon Signed-Rank test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons); p = 0.2437, Sign test — Wilcoxon Signed-Rank test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons)
Statistical Analysis 22: Comparison: Peer-led Intervention (PEER); [analysis description as in outcome 2, analysis 21]; Test type: Equivalence — Wilcoxon Signed-Rank test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons); p = 0.0631, Sign test — Wilcoxon Signed-Rank test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons)
Statistical Analysis 23: Comparison: Pharmacist-led Intervention (PHARM); Testing within-group changes in beliefs for the statement "I trust my pharmacist to give me information about vaccines and the diseases they prevent" from post-intervention to one-month follow-up; Test type: Equivalence — Wilcoxon Signed-Rank test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons); p = 0.0540, Sign test — Wilcoxon Signed-Rank test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons)
Statistical Analysis 24: Comparison: Peer-led Intervention (PEER); [analysis description as in outcome 2, analysis 23]; Test type: Equivalence — Wilcoxon Signed-Rank test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons); p = 0.7298, Sign test — Wilcoxon Signed-Rank test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons)
Statistical Analysis 25: Comparison: Pharmacist-led Intervention (PHARM); Testing within-group changes in beliefs for the statement "I trust a peer educator to give me information about vaccines and the diseases they prevent" from baseline to post-intervention; Test type: Equivalence — Wilcoxon Signed-Rank test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons); p = 0.4218, Sign test — Wilcoxon Signed-Rank test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons)
Statistical Analysis 26: Comparison: Peer-led Intervention (PEER); [analysis description as in outcome 2, analysis 25]; Test type: Equivalence — Wilcoxon Signed-Rank test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons); p = 0.2282, Sign test — Wilcoxon Signed-Rank test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons)
Statistical Analysis 27: Comparison: Pharmacist-led Intervention (PHARM); Testing within-group changes in beliefs for the statement "I trust a peer educator to give me information about vaccines and the diseases they prevent" from baseline to one-month follow-up; Test type: Equivalence — Wilcoxon Signed-Rank test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons); p = 0.8711, Sign test — Wilcoxon Signed-Rank test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons)
Statistical Analysis 28: Comparison: Peer-led Intervention (PEER); [analysis description as in outcome 2, analysis 27]; Test type: Equivalence — Wilcoxon Signed-Rank test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons); p = 0.0027, Sign test — Wilcoxon Signed-Rank test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons)
Statistical Analysis 29: Comparison: Pharmacist-led Intervention (PHARM); Testing within-group changes in beliefs for the statement "I trust a peer educator to give me information about vaccines and the diseases they prevent" from post-intervention to one-month follow-up; Test type: Equivalence — Wilcoxon Signed-Rank test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons); p = 0.7579, Sign test — Wilcoxon Signed-Rank test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons)
Statistical Analysis 30: Comparison: Peer-led Intervention (PEER); [analysis description as in outcome 2, analysis 29]; Test type: Equivalence — Wilcoxon Signed-Rank test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons); p = 0.1299, Sign test — Wilcoxon Signed-Rank test with a Bonferroni-corrected significance threshold of alpha = 0.0167 (3 comparisons)

3. Secondary Outcome: Cost Analysis
Description: Measure the program costs of PHARM and PEER from the senior center perspective. Costs were measured in total for each group, and per-participant costs were calculated by dividing total group cost by group sample size. Outcome measure type is thus reported as "number" rather than choosing measures of central tendency and dispersion/precision (i.e., there are no standard deviations, confidence intervals, or ranges with this methodology).
Time Frame: Measured after completion of all programs in both groups (an average of one year).
Measure: Number; unit: Dollars
Arm/Group | Pharmacist-led Intervention (PHARM) | Peer-led Intervention (PEER)
Number analyzed (Participants) | 147 | 140
Dollars
  Total cost in dollars | 7392.94 | 14887.45
  Total cost per participant | 50.29 | 106.34
  Total cost per session | 1232.16 | 1240.62
  Total senior center cost | 2488.98 | 5548.25
  Total senior center cost per participant | 16.93 | 39.63
  Staff cost (community health worker) | 417.49 | 1938.04
  Staff cost (PEER Leaders/Pharmacists) | 1109.14 | 1960.00
  Staff cost (Program Director) | 327.33 | 769.92
  Staff cost (Senior center director) | 0 | 281.24
  Total staff cost | 1853.96 | 4949.20
  Total staff cost per participant | 12.61 | 35.35
  Total staff cost per session | 308.99 | 412.43
  Travel costs | 378.89 | 342.92
  Space costs | 1500 | 3000
  Supplies cost | 256.13 | 256.13
  Refreshment costs | 1550.00 | 1390.00

4. Secondary Outcome: Number of Participants Reporting Program Satisfaction
Description: Satisfaction was assessed on the post-intervention and one-month follow-up surveys using two statements that were each scored on a 4-point Likert scale (1-Completely disagree, 2-Somewhat disagree, 3-Somewhat agree, 4-Completely agree). The statements were: 1) "The educational program kept me interested or engaged" and 2) "I was satisfied with the content of the educational program". At each timepoint, responses were dichotomized as "agree" (comprising the "Somewhat agree" and "Completely agree" response options) and "disagree" (comprising the "Somewhat disagree" and "Completely disagree" response options), and these dichotomous responses were compared between PHARM and PEER via Fisher's exact test.
Time Frame: Measured immediately post-intervention (PT) and at 1 month follow-up (1M)
Measure: Count of Participants; unit: Participants
Arm/Group | Pharmacist-led Intervention (PHARM) | Peer-led Intervention (PEER)
Number analyzed (Participants) | 147 | 140
Participants
  The program kept me interested or engaged - PT: Completely or somewhat agree | 124 | 127
  The program kept me interested or engaged - PT: Completely or somewhat disagree | 2 | 3
  The program kept me interested or engaged - PT: No response | 21 | 10
  The program kept me interested or engaged - 1M: Completely or somewhat agree | 130 | 135
  The program kept me interested or engaged - 1M: Completely or somewhat disagree | 3 | 2
  The program kept me interested or engaged - 1M: No response | 14 | 3
  I was satisfied with program content - PT: Completely or somewhat agree | 125 | 125
  I was satisfied with program content - PT: Completely or somewhat disagree | 1 | 2
  I was satisfied with program content - PT: No response | 21 | 13
  I was satisfied with program content - 1M: Completely or somewhat agree | 132 | 138
  I was satisfied with program content - 1M: Completely or somewhat disagree | 1 | 0
  I was satisfied with program content - 1M: No response | 14 | 2
Statistical Analysis 1: Comparison: Pharmacist-led Intervention (PHARM) vs Peer-led Intervention (PEER); Testing between-group differences in dichotomous engagement in the program immediately post-intervention via Fisher's Exact test; Test type: Equivalence — Fisher's Exact test was used (2 x 2) with a significance threshold of 0.05; p = 1.0, Fisher Exact — Fisher's Exact test was used (2 x 2) with a significance threshold of 0.05
Statistical Analysis 2: Comparison: Pharmacist-led Intervention (PHARM) vs Peer-led Intervention (PEER); Testing between-group differences in dichotomous engagement in the program at the one-month follow-up via Fisher's Exact test; Test type: Equivalence — Fisher's Exact test was used (2 x 2) with a significance threshold of 0.05; p = 0.6806, Fisher Exact — Fisher's Exact test was used (2 x 2) with a significance threshold of 0.05
Statistical Analysis 3: Comparison: Pharmacist-led Intervention (PHARM) vs Peer-led Intervention (PEER); Testing between-group differences in dichotomous satisfaction with the program's content immediately post-intervention via Fisher's Exact test; Test type: Equivalence — Fisher's Exact test was used (2 x 2) with a significance threshold of 0.05; p = 1.0, Fisher Exact — Fisher's Exact test was used (2 x 2) with a significance threshold of 0.05
Statistical Analysis 4: Comparison: Pharmacist-led Intervention (PHARM) vs Peer-led Intervention (PEER); Testing between-group differences in dichotomous satisfaction with the program's content at the one-month follow-up via Fisher's Exact test; Test type: Equivalence — Fisher's Exact test was used (2 x 2) with a significance threshold of 0.05; p = 0.4908, Fisher Exact — Fisher's Exact test was used (2 x 2) with a significance threshold of 0.05

5. Secondary Outcome: Number of Participants Planning to Receive Each Vaccine
Description: Compare the number of participants planning to receive vaccine in PHARM vs. PEER at each timepoint as assessed by the activation questionnaire
Time Frame: Measured at baseline (BL), immediately post-intervention (PT), and 1 month follow-up (1M)
Population: Rows labeled "Those without history of [...] vaccine" contain a subgroup analysis of those participants not reporting a positive vaccination history at post-test.
Measure: Count of Participants; unit: Participants
Arm/Group | Pharmacist-led Intervention (PHARM) | Peer-led Intervention (PEER)
Number analyzed (Participants) | 147 | 140
Participants
  Planning to receive zoster vaccine at BL: Planning to receive vaccine | 26 | 36
  Planning to receive zoster vaccine at BL: Not planning to receive vaccine | 46 | 58
  Planning to receive zoster vaccine at BL: No response | 75 | 46
  Planning to receive zoster vaccine at PT: Planning to receive vaccine | 44 | 60
  Planning to receive zoster vaccine at PT: Not planning to receive vaccine | 38 | 46
  Planning to receive zoster vaccine at PT: No response | 65 | 34
  Planning to receive zoster vaccine at 1M: Planning to receive vaccine | 46 | 56
  Planning to receive zoster vaccine at 1M: Not planning to receive vaccine | 44 | 57
  Planning to receive zoster vaccine at 1M: No response | 57 | 27
  Planning to receive influenza vaccine at BL: Planning to receive vaccine | 22 | 30
  Planning to receive influenza vaccine at BL: Not planning to receive vaccine | 25 | 36
  Planning to receive influenza vaccine at BL: No response | 100 | 74
  Planning to receive influenza vaccine at PT: Planning to receive vaccine | 35 | 44
  Planning to receive influenza vaccine at PT: Not planning to receive vaccine | 26 | 30
  Planning to receive influenza vaccine at PT: No response | 86 | 66
  Planning to receive influenza vaccine at 1M: Planning to receive vaccine | 36 | 45
  Planning to receive influenza vaccine at 1M: Not planning to receive vaccine | 27 | 36
  Planning to receive influenza vaccine at 1M: No response | 84 | 59
  Planning to receive pneumonia vaccine at BL: Planning to receive vaccine | 26 | 35
  Planning to receive pneumonia vaccine at BL: Not planning to receive vaccine | 35 | 35
  Planning to receive pneumonia vaccine at BL: No response | 86 | 70
  Planning to receive pneumonia vaccine at PT: Planning to receive vaccine | 40 | 55
  Planning to receive pneumonia vaccine at PT: Not planning to receive vaccine | 32 | 28
  Planning to receive pneumonia vaccine at PT: No response | 75 | 57
  Planning to receive pneumonia vaccine at 1M: Planning to receive vaccine | 45 | 54
  Planning to receive pneumonia vaccine at 1M: Not planning to receive vaccine | 37 | 40
  Planning to receive pneumonia vaccine at 1M: No response | 65 | 46
  Those without history of zoster vaccine (PT): number analyzed (Participants) | 93 | 110
  Those without history of zoster vaccine (PT): Planning to receive vaccine | 42 | 59
  Those without history of zoster vaccine (PT): Not planning to receive vaccine | 37 | 45
  Those without history of zoster vaccine (PT): No response | 14 | 6
  Those without history of zoster vaccine (1M): number analyzed (Participants) | 93 | 110
  Those without history of zoster vaccine (1M): Planning to receive vaccine | 39 | 53
  Those without history of zoster vaccine (1M): Not planning to receive vaccine | 43 | 54
  Those without history of zoster vaccine (1M): No response | 11 | 3
  Those without history of influenza vaccine (PT): number analyzed (Participants) | 61 | 69
  Those without history of influenza vaccine (PT): Planning to receive vaccine | 32 | 40
  Those without history of influenza vaccine (PT): Not planning to receive vaccine | 26 | 28
  Those without history of influenza vaccine (PT): No response | 3 | 1
  Those without history of influenza vaccine (1M): number analyzed (Participants) | 61 | 69
  Those without history of influenza vaccine (1M): Planning to receive vaccine | 31 | 38
  Those without history of influenza vaccine (1M): Not planning to receive vaccine | 27 | 31
  Those without history of influenza vaccine (1M): No response | 3 | 0
  Those without history of pneumonia vaccine (PT): number analyzed (Participants) | 75 | 71
  Those without history of pneumonia vaccine (PT): Planning to receive vaccine | 35 | 43
  Those without history of pneumonia vaccine (PT): Not planning to receive vaccine | 29 | 25
  Those without history of pneumonia vaccine (PT): No response | 11 | 3
  Those without history of pneumonia vaccine (1M): number analyzed (Participants) | 75 | 71
  Those without history of pneumonia vaccine (1M): Planning to receive vaccine | 34 | 36
  Those without history of pneumonia vaccine (1M): Not planning to receive vaccine | 33 | 32
  Those without history of pneumonia vaccine (1M): No response | 8 | 3
Statistical Analysis 1: Comparison: Pharmacist-led Intervention (PHARM) vs Peer-led Intervention (PEER); Testing between-group differences in number of participants planning to receive zoster vaccine at baseline via Chi-squared test; Test type: Equivalence — Chi-squared test was used with a significance threshold of 0.05; p = 0.7728, Chi-squared
Statistical Analysis 2: Comparison: Pharmacist-led Intervention (PHARM) vs Peer-led Intervention (PEER); Testing between-group differences in number of participants planning to receive zoster vaccine post-intervention via Chi-squared test; Test type: Equivalence — Chi-squared test was used with a significance threshold of 0.05; p = 0.6871, Chi-squared
Statistical Analysis 3: Comparison: Pharmacist-led Intervention (PHARM) vs Peer-led Intervention (PEER); Testing between-group differences in number of participants planning to receive zoster vaccine at one-month follow-up via Chi-squared test; Test type: Equivalence — Chi-squared test was used with a significance threshold of 0.05; p = 0.8259, Chi-squared
Statistical Analysis 4: Comparison: Pharmacist-led Intervention (PHARM) vs Peer-led Intervention (PEER); Testing between-group differences in number of participants planning to receive influenza vaccine at baseline via Chi-squared test; Test type: Equivalence — Chi-squared test was used with a significance threshold of 0.05; p = 0.8868, Chi-squared
Statistical Analysis 5: Comparison: Pharmacist-led Intervention (PHARM) vs Peer-led Intervention (PEER); Testing between-group differences in number of participants planning to receive influenza vaccine post-intervention via Chi-squared test; Test type: Equivalence — Chi-squared test was used with a significance threshold of 0.05; p = 0.8069, Chi-squared
Statistical Analysis 6: Comparison: Pharmacist-led Intervention (PHARM) vs Peer-led Intervention (PEER); Testing between-group differences in number of participants planning to receive influenza vaccine at one-month follow-up via Chi-squared test; Test type: Equivalence — Chi-squared test was used with a significance threshold of 0.05; p = 0.8489, Chi-squared
Statistical Analysis 7: Comparison: Pharmacist-led Intervention (PHARM) vs Peer-led Intervention (PEER); Testing between-group differences in number of participants planning to receive pneumonia vaccine at baseline via Chi-squared test; Test type: Equivalence — Chi-squared test was used with a significance threshold of 0.05; p = 0.3985, Chi-squared
Statistical Analysis 8: Comparison: Pharmacist-led Intervention (PHARM) vs Peer-led Intervention (PEER); Testing between-group differences in number of participants planning to receive pneumonia vaccine post-intervention via Chi-squared test; Test type: Equivalence — Chi-squared test was used with a significance threshold of 0.05; p = 0.1722, Chi-squared
Statistical Analysis 9: Comparison: Pharmacist-led Intervention (PHARM) vs Peer-led Intervention (PEER); Testing between-group differences in number of participants planning to receive pneumonia vaccine at one-month follow-up via Chi-squared test; Test type: Equivalence — Chi-squared test was used with a significance threshold of 0.05; p = 0.7318, Chi-squared
Statistical Analysis 10: Comparison: Pharmacist-led Intervention (PHARM) vs Peer-led Intervention (PEER); Among those without positive vaccination history at post-test, testing between-group differences in number of participants planning to receive zoster vaccine post-intervention via Chi-squared test; Test type: Equivalence — Chi-squared test was used with a significance threshold of 0.05; p = 0.6309, Chi-squared
Statistical Analysis 11: Comparison: Pharmacist-led Intervention (PHARM) vs Peer-led Intervention (PEER); Among those without positive vaccination history at post-test, testing between-group differences in number of participants planning to receive zoster vaccine at one-month follow-up via Chi-squared test; Test type: Equivalence — Chi-squared test was used with a significance threshold of 0.05; p = 0.7881, Chi-squared
Statistical Analysis 12: Comparison: Pharmacist-led Intervention (PHARM) vs Peer-led Intervention (PEER); Among those without positive vaccination history at post-test, testing between-group differences in number of participants planning to receive influenza vaccine post-intervention via Chi-squared test; Test type: Equivalence — Chi-squared test was used with a significance threshold of 0.05; p = 0.6798, Chi-squared
Statistical Analysis 13: Comparison: Pharmacist-led Intervention (PHARM) vs Peer-led Intervention (PEER); Among those without positive vaccination history at post-test, testing between-group differences in number of participants planning to receive influenza vaccine at one-month follow-up via Chi-squared test; Test type: Equivalence — Chi-squared test was used with a significance threshold of 0.05; p = 0.8548, Chi-squared
Statistical Analysis 14: Comparison: Pharmacist-led Intervention (PHARM) vs Peer-led Intervention (PEER); Among those without positive vaccination history at post-test, testing between-group differences in number of participants planning to receive pneumonia vaccine post-intervention via Chi-squared test; Test type: Equivalence — Chi-squared test was used with a significance threshold of 0.05; p = 0.3182, Chi-squared
Statistical Analysis 15: Comparison: Pharmacist-led Intervention (PHARM) vs Peer-led Intervention (PEER); Among those without positive vaccination history at post-test, testing between-group differences in number of participants planning to receive pneumonia vaccine at one-month follow-up via Chi-squared test; Test type: Equivalence — Chi-squared test was used with a significance threshold of 0.05; p = 0.7986, Chi-squared

6. Secondary Outcome: Number of Participants Reporting Positive Vaccination Status at Each Timepoint
Description: Compare the number participants reporting positive vaccination status in PHARM vs. PEER at each timepoint as assessed by the activation questionnaire
Time Frame: Measured at baseline (BL), immediately post-intervention (PT), and 1 month follow-up (1M)
Population: Rows labeled "without previous [...] vaccine", contain a subgroup analysis of those participants not reporting a positive vaccination history at post-test.
Measure: Count of Participants; unit: Participants
Arm/Group | Pharmacist-led Intervention (PHARM) | Peer-led Intervention (PEER)
Number analyzed (Participants) | 147 | 140
Participants
  Reporting history of zoster vaccine at BL: Yes | 50 | 32
  Reporting history of zoster vaccine at BL: No | 80 | 98
  Reporting history of zoster vaccine at BL: No response | 17 | 10
  Reporting history of zoster vaccine at PT: Yes | 54 | 30
  Reporting history of zoster vaccine at PT: No | 85 | 105
  Reporting history of zoster vaccine at PT: No response | 8 | 5
  Reporting history of zoster vaccine at 1M: Yes | 52 | 36
  Reporting history of zoster vaccine at 1M: No | 88 | 103
  Reporting history of zoster vaccine at 1M: No response | 7 | 1
  Reporting history of influenza vaccine at BL: Yes | 86 | 70
  Reporting history of influenza vaccine at BL: No | 51 | 66
  Reporting history of influenza vaccine at BL: No response | 10 | 4
  Reporting history of influenza vaccine at PT: Yes | 86 | 71
  Reporting history of influenza vaccine at PT: No | 60 | 68
  Reporting history of influenza vaccine at PT: No response | 1 | 1
  Reporting history of influenza vaccine at 1M: Yes | 89 | 81
  Reporting history of influenza vaccine at 1M: No | 57 | 59
  Reporting history of influenza vaccine at 1M: No response | 1 | 0
  Reporting history of pneumonia vaccine at BL: Yes | 65 | 59
  Reporting history of pneumonia vaccine at BL: No | 67 | 75
  Reporting history of pneumonia vaccine at BL: No response | 15 | 6
  Reporting history of pneumonia vaccine at PT: Yes | 72 | 69
  Reporting history of pneumonia vaccine at PT: No | 70 | 69
  Reporting history of pneumonia vaccine at PT: No response | 5 | 2
  Reporting history of pneumonia vaccine at 1M: Yes | 69 | 67
  Reporting history of pneumonia vaccine at 1M: No | 75 | 72
  Reporting history of pneumonia vaccine at 1M: No response | 3 | 1
  Those without zoster vaccine at PT (1M status): number analyzed (Participants) | 93 | 110
  Those without zoster vaccine at PT (1M status): Yes | 3 | 10
  Those without zoster vaccine at PT (1M status): No | 83 | 99
  Those without zoster vaccine at PT (1M status): No response | 7 | 1
  Those without influenza vaccine at PT (1M status): number analyzed (Participants) | 61 | 69
  Those without influenza vaccine at PT (1M status): Yes | 5 | 17
  Those without influenza vaccine at PT (1M status): No | 55 | 52
  Those without influenza vaccine at PT (1M status): No response | 1 | 0
  Those without pneumonia vaccine at PT (1M status): number analyzed (Participants) | 75 | 71
  Those without pneumonia vaccine at PT (1M status): Yes | 6 | 14
  Those without pneumonia vaccine at PT (1M status): No | 66 | 56
  Those without pneumonia vaccine at PT (1M status): No response | 3 | 1
Statistical Analysis 1: Comparison: Pharmacist-led Intervention (PHARM) vs Peer-led Intervention (PEER); Testing between-group differences in number of participants reporting positive history of zoster vaccine at baseline via Chi-squared test; Test type: Equivalence — Chi-squared test was used with a significance threshold of 0.05; p = 0.0163, Chi-squared
Statistical Analysis 2: Comparison: Pharmacist-led Intervention (PHARM) vs Peer-led Intervention (PEER); Testing between-group differences in number of participants reporting positive history of zoster vaccine post-intervention via Chi-squared test; Test type: Equivalence — Chi-squared test was used with a significance threshold of 0.05; p = 0.0028, Chi-squared
Statistical Analysis 3: Comparison: Pharmacist-led Intervention (PHARM) vs Peer-led Intervention (PEER); Testing between-group differences in number of participants reporting positive history of zoster vaccine at one-month follow-up via Chi-squared test; Test type: Equivalence — Chi-squared test was used with a significance threshold of 0.05; p = 0.0433, Chi-squared
Statistical Analysis 4: Comparison: Pharmacist-led Intervention (PHARM) vs Peer-led Intervention (PEER); Testing between-group differences in number of participants reporting positive history of influenza vaccine at baseline via Chi-squared test; Test type: Equivalence — Chi-squared test was used with a significance threshold of 0.05; p = 0.0592, Chi-squared
Statistical Analysis 5: Comparison: Pharmacist-led Intervention (PHARM) vs Peer-led Intervention (PEER); Testing between-group differences in number of participants reporting positive history of influenza vaccine post-intervention via Chi-squared test; Test type: Equivalence — Chi-squared test was used with a significance threshold of 0.05; p = 0.1843, Chi-squared
Statistical Analysis 6: Comparison: Pharmacist-led Intervention (PHARM) vs Peer-led Intervention (PEER); Testing between-group differences in number of participants reporting positive history of influenza vaccine at one-month follow-up via Chi-squared test; Test type: Equivalence — Chi-squared test was used with a significance threshold of 0.05; p = 0.5933, Chi-squared
Statistical Analysis 7: Comparison: Pharmacist-led Intervention (PHARM) vs Peer-led Intervention (PEER); Testing between-group differences in number of participants reporting positive history of pneumonia vaccine at baseline via Chi-squared test; Test type: Equivalence — Chi-squared test was used with a significance threshold of 0.05; p = 0.3942, Chi-squared
Statistical Analysis 8: Comparison: Pharmacist-led Intervention (PHARM) vs Peer-led Intervention (PEER); Testing between-group differences in number of participants reporting positive history of pneumonia vaccine post-intervention via Chi-squared test; Test type: Equivalence — Chi-squared test was used with a significance threshold of 0.05; p = 0.9062, Chi-squared
Statistical Analysis 9: Comparison: Pharmacist-led Intervention (PHARM) vs Peer-led Intervention (PEER); Testing between-group differences in number of participants reporting positive history of pneumonia vaccine at one-month follow-up via Chi-squared test; Test type: Equivalence — Chi-squared test was used with a significance threshold of 0.05; p = 0.9618, Chi-squared
Statistical Analysis 10: Comparison: Pharmacist-led Intervention (PHARM) vs Peer-led Intervention (PEER); Among those without positive vaccination history at post-test, testing between-group differences in number of participants reporting positive history of zoster vaccine at one-month follow-up via Chi-squared test; Test type: Equivalence — Chi-squared test was used with a significance threshold of 0.05; p = 0.1140, Chi-squared
Statistical Analysis 11: Comparison: Pharmacist-led Intervention (PHARM) vs Peer-led Intervention (PEER); Among those without positive vaccination history at post-test, testing between-group differences in number of participants reporting positive history of influenza vaccine at one-month follow-up via Chi-squared test; Test type: Equivalence — Chi-squared test was used with a significance threshold of 0.05; p = 0.0141, Chi-squared
Statistical Analysis 12: Comparison: Pharmacist-led Intervention (PHARM) vs Peer-led Intervention (PEER); Among those without positive vaccination history at post-test, testing between-group differences in number of participants reporting positive history of pneumonia vaccine at one-month follow-up via Chi-squared test; Test type: Equivalence — Chi-squared test was used with a significance threshold of 0.05; p = 0.0457, Chi-squared

7. Secondary Outcome: Number of Participants Planning to Discuss Vaccines With Others as Assessed by the Activation Questionnaire
Description: Compare the number of participants planning to discuss vaccines with doctor, pharmacist, or family/friends in PHARM vs. PEER at each timepoint
Time Frame: Baseline, immediately post-intervention, and 1 month follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Pharmacist-led Intervention (PHARM) | Peer-led Intervention (PEER)
Number analyzed (Participants) | 147 | 140
Participants
  Planning to discuss with doctor at BL: Yes | 66 | 67
  Planning to discuss with doctor at BL: No response | 81 | 73
  Planning to discuss with doctor at PT: Yes | 98 | 95
  Planning to discuss with doctor at PT: No response | 49 | 45
  Planning to discuss with doctor at 1M: Yes | 112 | 120
  Planning to discuss with doctor at 1M: No response | 35 | 20
  Planning to discuss with pharmacist at BL: Yes | 15 | 19
  Planning to discuss with pharmacist at BL: No response | 132 | 121
  Planning to discuss with pharmacist at PT: Yes | 30 | 36
  Planning to discuss with pharmacist at PT: No response | 117 | 104
  Planning to discuss with pharmacist at 1M: Yes | 38 | 61
  Planning to discuss with pharmacist at 1M: No response | 109 | 79
  Planning to discuss with family/friends at BL: Yes | 14 | 13
  Planning to discuss with family/friends at BL: No response | 133 | 127
  Planning to discuss with family/friends at PT: Yes | 30 | 32
  Planning to discuss with family/friends at PT: No response | 117 | 108
  Planning to discuss with family/friends at 1M: Yes | 39 | 60
  Planning to discuss with family/friends at 1M: No response | 108 | 80
Statistical Analysis 1: Comparison: Pharmacist-led Intervention (PHARM) vs Peer-led Intervention (PEER); Testing between-group differences in number of participants planning to discuss vaccines with their doctor at baseline via Chi-squared test; Test type: Equivalence — Chi-squared test was used with a significance threshold of 0.05; p = 0.6153, Chi-squared
Statistical Analysis 2: Comparison: Pharmacist-led Intervention (PHARM) vs Peer-led Intervention (PEER); Testing between-group differences in number of participants planning to discuss vaccines with their doctor post-intervention via Chi-squared test; Test type: Equivalence — Chi-squared test was used with a significance threshold of 0.05; p = 0.8299, Chi-squared
Statistical Analysis 3: Comparison: Pharmacist-led Intervention (PHARM) vs Peer-led Intervention (PEER); Testing between-group differences in number of participants planning to discuss vaccines with their doctor at one-month follow-up via Chi-squared test; Test type: Equivalence — Chi-squared test was used with a significance threshold of 0.05; p = 0.0405, Chi-squared
Statistical Analysis 4: Comparison: Pharmacist-led Intervention (PHARM) vs Peer-led Intervention (PEER); Testing between-group differences in number of participants planning to discuss vaccines with their pharmacist at baseline via Chi-squared test; Test type: Equivalence — Chi-squared test was used with a significance threshold of 0.05; p = 0.3776, Chi-squared
Statistical Analysis 5: Comparison: Pharmacist-led Intervention (PHARM) vs Peer-led Intervention (PEER); Testing between-group differences in number of participants planning to discuss vaccines with their pharmacist post-intervention via Chi-squared test; Test type: Equivalence — Chi-squared test was used with a significance threshold of 0.05; p = 0.2856, Chi-squared
Statistical Analysis 6: Comparison: Pharmacist-led Intervention (PHARM) vs Peer-led Intervention (PEER); Testing between-group differences in number of participants planning to discuss vaccines with their pharmacist at one-month follow-up via Chi-squared test; Test type: Equivalence — Chi-squared test was used with a significance threshold of 0.05; p = 0.0016, Chi-squared
Statistical Analysis 7: Comparison: Pharmacist-led Intervention (PHARM) vs Peer-led Intervention (PEER); Testing between-group differences in number of participants planning to discuss vaccines with their family/friends at baseline via Chi-squared test; Test type: Equivalence — Chi-squared test was used with a significance threshold of 0.05; p = 0.9449, Chi-squared
Statistical Analysis 8: Comparison: Pharmacist-led Intervention (PHARM) vs Peer-led Intervention (PEER); Testing between-group differences in number of participants planning to discuss vaccines with their family/friends post-intervention via Chi-squared test; Test type: Equivalence — Chi-squared test was used with a significance threshold of 0.05; p = 0.6143, Chi-squared
Statistical Analysis 9: Comparison: Pharmacist-led Intervention (PHARM) vs Peer-led Intervention (PEER); Testing between-group differences in number of participants planning to discuss vaccines with their family/friends at one-month follow-up via Chi-squared test; Test type: Equivalence — Chi-squared test was used with a significance threshold of 0.05; p = 0.0036, Chi-squared

8. Secondary Outcome: Number of Participants Having Discussed Vaccines With Others at One-month Follow-up as Assessed by the Activation Questionnaire
Description: Compare the number of participants reporting that they have discussed vaccines with their doctor, pharmacist, or family/friends at the one-month follow-up for PHARM vs. PEER
Time Frame: One-month follow-up (1M)
Measure: Count of Participants; unit: Participants
Arm/Group | Pharmacist-led Intervention (PHARM) | Peer-led Intervention (PEER)
Number analyzed (Participants) | 147 | 140
Participants
  Discussed with doctor at 1M: Yes | 22 | 62
  Discussed with doctor at 1M: No response | 125 | 78
  Discussed with pharmacist at 1M: Yes | 7 | 23
  Discussed with pharmacist at 1M: No response | 140 | 117
  Discussed with family/friends at 1M: Yes | 9 | 24
  Discussed with family/friends at 1M: No response | 138 | 116
Statistical Analysis 1: Comparison: Pharmacist-led Intervention (PHARM) vs Peer-led Intervention (PEER); Testing between-group differences in number of participants having discussed vaccines with their doctor at one-month follow-up via Chi-squared test; Test type: Equivalence — Chi-squared test was used with a significance threshold of 0.05; p < 0.0001, Chi-squared
Statistical Analysis 2: Comparison: Pharmacist-led Intervention (PHARM) vs Peer-led Intervention (PEER); Testing between-group differences in number of participants having discussed vaccines with their pharmacist at one-month follow-up via Chi-squared test; Test type: Equivalence — Chi-squared test was used with a significance threshold of 0.05; p = 0.0012, Chi-squared
Statistical Analysis 3: Comparison: Pharmacist-led Intervention (PHARM) vs Peer-led Intervention (PEER); Testing between-group differences in number of participants having discussed vaccines with their family/friends at one-month follow-up via Chi-squared test; Test type: Equivalence — Chi-squared test was used with a significance threshold of 0.05; p = 0.0034, Chi-squared

ADVERSE EVENTS:
Time Frame: Not Applicable - Study was a minimal-risk educational intervention.
Description: The study was an educational intervention deemed to present minimal risk to subjects. No adverse events were possible with this study. All-cause mortality, serious and other (not including serious) adverse events were not monitored.
Arm/Group | Pharmacist-led Intervention (PHARM) | Peer-led Intervention (PEER)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Study results may not be generalizable to non-Black subpopulations. Real number receiving the vaccination could be either higher or lower than reported due to self-report. Peer leader trust might have already been established prior to the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-05-01): https://cdn.clinicaltrials.gov/large-docs/65/NCT03239665/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-06): https://cdn.clinicaltrials.gov/large-docs/65/NCT03239665/SAP_001.pdf